CLINICAL TRIAL: NCT05454761
Title: Effects of Multicomponent Lifestyle Intervention for Depression Supported With Digital Health Technologies to Promote Adherence: A Randomized Controlled Trial and a Process Evaluation
Brief Title: Multicomponent Lifestyle Intervention for Depression Supported With Digital Health Technologies to Promote Adherence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Fiona YY Ho, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSY022
Record Dates: First submitted 2022-07-08; First posted 2022-07-12 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Depression
Keywords: Lifestyle Medicine; Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lifestyle medicine intervention with self-tracking tools (Experimental): Lifestyle intervention including diet, sleep, exercise, relaxation, and mindfulness. Self-tracking tools including a smartphone application and an Actigraphy will be given.
  Interventions: Behavioral: Group-based Lifestyle Medicine Program
- Pure lifestyle medicine intervention (Experimental): Lifestyle intervention including diet, sleep, exercise, relaxation, and mindfulness.
  Interventions: Behavioral: Group-based Lifestyle Medicine Program
- Care-As-Usual (No Intervention): continue receiving the routine care as usual and be given a smartphone-based LM intervention after the completion of follow-up assessments

INTERVENTIONS:
Behavioral: Group-based Lifestyle Medicine Program — Participants will receive four core modules that focus on lifestyle modifications. Core Module 1 will be Diets and Nutrition. This module aims to provide simple and evidence-based information regarding nutrition for improving and maintaining mental health. Core Module 2 will be Physical Activity. Participants will practice various types of gentle and adaptable exercises during the session and learn simple ways to incorporate exercise into their daily lives. Core Module 3 will be Sleep Management. This module will include basic facts about sleep, with a focus on psychoeducation on insomnia and how the relationship between circadian and social rhythms relate to sleep and mental health. Core Module 4 will be Stress Management. This module will include psychoeducation about stress, worry management, the cultivation of positive psychology, and relaxation techniques such as diaphragmatic breathing and progressive muscle relaxation.
  Arms: Lifestyle medicine intervention with self-tracking tools; Pure lifestyle medicine intervention

SUMMARY:
The proposed study will be a randomized, assessor-blind controlled trial embedding both outcome and process evaluations of a 6-week group LM intervention with/without self-tracking tools (Study I). The outcome evaluation will examine the effects of LM-S and LM alone vs. CAU, and the process evaluation will enhance the understanding of the causal assumptions that underpin LM to inform policy and clinical practice. Eligible participants with at least a moderate level of depression will be randomly assigned to the LM- S, LM alone, and CAU groups in a 1:1:1 allocation ratio. The study period will be 18 weeks. Assessments at baseline, week 7 (1-week post-intervention), and week 18 (12-week post-intervention) will be managed by an independent assessor (a research assistant, RA) who is blind to the group allocation. The proposed trial and the nested pilot study will follow the CONSORT and STROBE guidelines, respectively. The intervention will be provided free of charge.

ELIGIBILITY:
Inclusion Criteria:

1. at least 18 years of age
2. Cantonese language fluency and readability
3. a PHQ-9 score of at least 10, indicating a moderate level of depression
4. current DSM-IV diagnostic criteria of major depressive episode based on the Mini International Neuropsychiatric Interview (MINI)
5. possession of an internet-enabled mobile device (iOS or Android operating system)
6. willingness to provide informed consent and comply with the trial protocol.

Exclusion Criteria:

1. the presence of other current psychiatric disorders as assessed by the MINI
2. any medical or neurocognitive disorder(s) that makes participation unsuitable based on the team's clinical experience or interferes with adherence to the lifestyle modification (e.g., where exercise or a change in diet are not recommended by physicians)
3. current serious suicidal risk (non-fleeting intent or plan) as assessed by a PHQ-9 Item 9 score > 2 (referral information to professional mental health services will be provided)
4. current involvement in lifestyle changes supervised by professionals
5. intake of medication or current participation in any psychotherapy for depression
6. pregnancy
7. hospitalization
8. current participation in any other trial(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in the Patient Health Questionnaire (PHQ-9) | [Time Frame: Baseline, immediately after treatment, and 12 weeks after the treatment sessions are completed]
  The PHQ-9, a 20-item questionnaire used for screening, diagnosing, monitoring and measuring the severity of depression, which scores each of the nine DSM-IV criteria as "0" (not at all) to "3" (nearly every day).

SECONDARY OUTCOMES:
Change in Insomnia Severity Index (ISI) | [Time Frame: Baseline, immediately after treatment, and 12 weeks after the treatment sessions are completed]
  ISI is a 7-item scale designed to evaluate perceived insomnia severity. Ratings on the 5-point Likert scale are obtained on the perceived severity of sleep-onset, sleep-maintenance, early morning awakening problems, satisfaction with current sleep pattern, interference with daily functioning, noticeably of impairment attributed to the sleep problem, and level of distress caused by the sleep problem.
Change in the Health-Promoting Lifestyle Profile (HPLP II) | [Time Frame: Baseline, immediately after treatment, and 12 weeks after the treatment sessions are completed]
  The 52-item HPLPII is composed of a total scale and six subscales to measure behaviors in the theorized dimensions of health-promoting lifestyle: spiritual growth, interpersonal relations, nutrition, physical activity, health responsibility, and stress management.
Change in the Sheehan Disability Scale (SDS) | [Time Frame: Baseline, immediately after treatment, and 12 weeks after the treatment sessions are completed]
  SDS is a brief, 5-item self-report tool that assesses functional impairment in work/school, social life, and family life
Change in Quality-adjusted Life Years - The Short Form Six-Dimension (SF-6D) | [Time Frame: Baseline, immediately after treatment, and 12 weeks after the treatment sessions are completed]
  The Short Form Six-Dimension (SF-6D) is a self-report measure that assesses health-related quality of life to estimate participant's quality-adjusted life years (QALYs). This instrument was validated in the Chinese population and widely applied in previous mental health research.
Change in Hospital Anxiety and Depression Scale (HADS) | [Time Frame: Baseline, immediately after treatment, and 12 weeks after the treatment sessions are completed]
  HADS is a 14-item self-rated questionnaire which consists of two 7-item subscales that measure the presence of anxiety and depression symptoms respectively. Each item is rated on a 4-point-scale (0-3) by the participant. The greater the score, the more psychologically distressed the respondent is.

OTHER OUTCOMES:
Change in the Credibility-Expectancy Questionnaire (CEQ) | [Time Frame: Baseline and immediately after treatment]
  The 6-item CEQ yielded ratings of treatment credibility, acceptability/satisfaction, and expectations for success.
Treatment Acceptability Scale (TAS) | [Time Frame: Baseline and immediately after treatment]
  An 8-item scale of the willingness to utilize or recommend the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Shatin, Hong Kong